CLINICAL TRIAL: NCT01497314
Title: An Open Label Clinical Study to Evaluate Growth and Safety of a Low Lactose Milk-Based Infant Formula in Healthy Term Infants
Brief Title: Growth and Safety of a Low Lactose Milk-Based Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perrigo Nutritionals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PRG-VA-12-001
Record Dates: First submitted 2011-12-15; First posted 2011-12-22 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Growth; Healthy Term Infants
Keywords: healthy term infants; growth; infant formula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Lactose Infant Formula (Other)
  Interventions: Other: Low Lactose Infant Formula

INTERVENTIONS:
Other: Low Lactose Infant Formula — Low Lactose Infant Formula

SUMMARY:
The purpose of this study is to show that a low lactose milk-based infant formula supports normal growth in healthy term infants.

DETAILED DESCRIPTION:
Infants will be fed a low lactose milk-based formula for 16 weeks. Growth and formula tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy term infants
* birth weight 2500 - 4500 g
* singleton birth
* 37 - 42 weeks gestation

Exclusion Criteria:

* clinically significant abnormal findings (as determined by the investigator) on the physical examination or medical history
* receiving medications other than vitamins

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Weight | 16 weeks

SECONDARY OUTCOMES:
Length gain | 16 weeks
Occipital Head Circumference | 16 weeks
Acceptability and Tolerability | 16 weeks
  Assessed by digestive tolerance; general health and well-being; adverse events; concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Barber, PhD, Study Director — Perrigo Nutritionals
Locations (6):
- United States (6):
  - Accelovance Melbourne Site, Melbourne, Florida
  - ACC Pediatric Research, Haughton, Louisiana
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Research Across America, Dallas, Texas
  - Jean Brown Research, Murray, Utah
  - PI-Coor Research, Burke, Virginia